CLINICAL TRIAL: NCT06211491
Title: Autonomic Dysreflexia Clinical Characteristics According to the Filling Speed in Urodynamics in Individuals With Spinal Cord Injuries
Brief Title: Autonomic Dysreflexia in Spinal Cord Injuries: UDS Filling Speed Impact
Status: Recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sungchul Huh, Assistant Professor, Pusan National University Yangsan Hospital
Other Study IDs: UDS filling speed
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Autonomic Dysreflexia; UDS Filling Speed
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Urodynamic test — Urodynamic testing is performed using saline solution at the same temperature as body temperature (37 degrees) at two injection speeds of 10 mL/min and 100 mL/min, respectively.

SUMMARY:
In patients with spinal cord injury, the investigators want to understand and understand the differences in AD prevalence and characteristics according to bladder injection rate, and to determine which factors have a greater influence between bladder expansion or injection rate.

DETAILED DESCRIPTION:
It has been reported that there is a difference in the degree of AD between the bladder and urinary tract motility tests, suggesting a potential difference according to the injection rate. According to Liu et al., the authors noted that stimulation of the urethra, prostate, and internal sphincter appears to induce AD more strongly than the injection rate. In addition, the two main factors contributing to AD among urinary kinetics tests are the patient's age and bladder maximum urination pressure. Considering these factors is important in preventing AD during urinary kinetics tests. Despite these previous studies, the prevalence and severity of AD according to the injection rate of urinary kinetics tests in SCI have not been quantitatively evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic spinal cord injury 6 months after receiving the award
2. Patients with confirmed AD due to bladder fullness in previous urodynamic test
3. Patients confirmed to have neurological damage level C1-T6, AIS A or B

Exclusion Criteria:

1. Patients who cannot perform the test because their systolic blood pressure remains at 150 mmHg during the urodynamic test
2. Patients who cannot undergo testing due to hemodynamic instability
3. Patients who cannot undergo testing due to overt urinary tract infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic spinal cord injuries
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Bladder volume (ml) | Immediately after the test
  (1) at first AD at an infusion rate of 10 mL/min (2) at first AD at an infusion rate of 100 mL/min

SECONDARY OUTCOMES:
Bladder compliance (mL/cmH2O) | Immediately after the test
  Bladder compliance
Symptoms (Y/N) | Immediately after the test
  Symptoms
Blood pressure (mmHg) | Immediately after the test
  Blood pressure
Heart rate (bpm) | Immediately after the test
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Sungchul Huh, Ph.D, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No